CLINICAL TRIAL: NCT02211066
Title: TIcaGrEloR and ABSORB Bioresorbable Vascular Scaffold Implantation for Recovery of Vascular Function After Successful Chronic Total Occlusion Recanalization
Acronym: TIGER-BVS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Juan A. Arnaiz, Clinical Trial Manager, Hospital Clinic of Barcelona
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TIGER-BVS; 2013-002675-17 (EudraCT Number)
Record Dates: First submitted 2014-07-28; First posted 2014-08-07 (Estimated); Last update posted 2019-12-19 (Actual); Status verified 2019-12

CONDITIONS: Patients Who Are Scheduled to Undergo a PCI (Percutaneous Coronary Intervention) for CTO (Chronic Total Occlusion)
MeSH Terms: interventions — Clopidogrel; Ticagrelor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Clopidogrel (Active Comparator): Clopidogrel 75 mg will be administered daily for 1 year
  Interventions: Drug: Clopidogrel
- Ticagrelor (Experimental): Ticagrelor 90 mg will be administered daily for 1 year
  Interventions: Drug: Ticagrelor

INTERVENTIONS:
Drug: Clopidogrel
  Arms: Clopidogrel
Drug: Ticagrelor
  Arms: Ticagrelor

SUMMARY:
The study is a single-centre, randomized, active controlled, open label clinical trial. The primary hypothesis is that ticagrelor will show superiority over clopidogrel immediately after CTO-PCI (chronic total occlusion - percutaneous coronary intervention)

DETAILED DESCRIPTION:
The hypothesis is tested in the first randomization. Both antiplatelet therapy will be used in both arms at the approved doses and for the approved duration therapy of 1-year. The secondary hypothesis will test the role of ticagrelor/clopidogrel alone and together with ABSORB BVS implantation in the recovery of vascular function at long-term. This hypothesis is tested in the second randomization. The angiographic follow-up will be scheduled at 1 or 3-year follow-up in order to test the secondary hypothesis either at the moment of the end of the antiplatelet therapy or at the moment of scaffold bioresorption.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes, older than 18 years old.
* Written informed consent obtained.
* Patients with stable angina pectoris (Canadian Cardiovascular Society (CCS) Class 1, 2, 3 or 4) or patients with documented silent ischemia by stress test during the last year.
* Patients eligible for coronary revascularization in a coronary chronic total occlusion, which was angiographically documented in a previous coronary angiography during the last year.

Exclusion Criteria:

* Women who are pregnant or women of childbearing potential who do not use adequate contraception.
* Known allergies to aspirin, clopidogrel bisulfate (Plavix ®), ticagrelor (BriliqueTM) heparin, or a sensitivity to contrast media, which cannot be adequately pre-medicated.
* Participation in other studies.
* Life expectancy of less than one year or factors making clinical and/or angiographic follow-up difficult.
* Planned cardiac surgery or major non-cardiac surgery.
* The subject has a history of bleeding diathesis or coagulopathy.
* The subject suffered disabling stroke within the past year.
* Known major hematologic, neoplastic, metabolic, gastrointestinal or endocrine dysfunction, which, in the judgment of the Investigator, may affect the patient's ability to complete the study.
* History of malignancy, except in patients who have been disease-free >5 years or whose only malignancy has been basal or squamous cell skin carcinoma.
* Inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2014-10; Primary Completion 2019-06 (Actual); Study Completion 2019-06-12 (Actual)

PRIMARY OUTCOMES:
Differences in increase of coronary blood flow (CBF) under adenosine administration from baseline in the coronary segment distal to the scaffold implanted immediately after CTO-PCI between the ticagrelor vs. clopidogrel group. | Baseline

SECONDARY OUTCOMES:
Changes from baseline in mean lumen diameter after nitrate administration in the coronary segment distal to the scaffold implanted immediately after CTO-PCI between the ticagrelor vs. clopidogrel group. | Baseline
Changes from baseline in coronary flow reserve after adenosine administration in the coronary segment distal to the scaffold implanted immediately after CTO-PCI between the ticagrelor vs. clopidogrel group. | Baseline
Changes from baseline in mean lumen diameter after nitrate administration in the coronary segment scaffolded by ABSORB and in that distal to it at 1 year follow-up between the ticagrelor vs. clopidogrel group. | 1 year
Changes from baseline in coronary blood flow after adenosine administration in the coronary segment distal to the scaffold implanted at 1-year follow-up between the ticagrelor vs. clopidogrel group | 1 year
Changes from baseline in coronary flow reserve after adenosine administration in the coronary segment distal to the scaffold implanted at 1-year follow-up between the ticagrelor vs. clopidogrel group. | 1 year
Changes from baseline in mean lumen diameter after nitrate administration in the coronary segment scaffolded by ABSORB and in that distal to it at 3-year follow-up between the ticagrelor vs. clopidogrel group. | 3 years
Changes from baseline in coronary blood flow after adenosine administration in the coronary segment distal to the scaffold implanted at 3-year follow-up between the ticagrelor vs. clopidogrel group. | 3 years
Changes from baseline in coronary flow reserve after adenosine administration in the coronary segment distal to the scaffold implanted at 3-year follow-up between the ticagrelor vs. clopidogrel group. | 3 years
Difference in intimal-media thickness at the site of scaffold implanted, evaluated by optical coherence tomography in a subgroup of patients at 1-year follow-up between the ticagrelor vs. clopidogrel group. | 1 year
Difference in intimal-media thickness at the site of scaffold implanted, evaluated by optical coherence tomography at 3 years follow-up between the ticagrelor vs. clopidogrel group. | 3 years
Clinical endpoints at 1 and 3 years follow-up: cardiac death, probable or definite scaffold thrombosis, target vessel failure, bleeding. | 1 and 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Salvatore Brugaletta, MD, Principal Investigator — Hospital Clinic of Barcelona
Locations (2):
- Spain (2):
  - Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital Clínic de Barcelona, Barcelona

REFERENCES:
- [Derived] Rodriguez-Arias JJ, Gomez-Lara J, Caballero-Borrego J, Ortega-Paz L, Arevalos V, Teruel L, Gil-Jimenez T, Oyarzabal L, Romaguera R, Moreno-Terribas G, Gomez-Hospital JA, Sabate M, Brugaletta S. Long-Term Vascular Function in CTO Recanalization: A Randomized Clinical Trial of Ticagrelor vs. Clopidogrel. Cardiovasc Revasc Med. 2022 Apr;37:61-67. doi: 10.1016/j.carrev.2021.06.129. Epub 2021 Jul 1. PMID 34238679
- [Derived] Brugaletta S, Gomez-Lara J, Caballero J, Ortega-Paz L, Teruel L, Jimenez Fernandez M, Romaguera R, Alcalde Martinez V, Nato M, Molina Navarro E, Gomez-Hospital JA, Correa Vilches C, Joyera M, Cequier A, Sabate M. TIcaGrEloR and Absorb bioresorbable vascular scaffold implantation for recovery of vascular function after successful chronic total occlusion recanalization (TIGER-BVS trial): Rationale and study design. Catheter Cardiovasc Interv. 2018 Jan 1;91(1):1-6. doi: 10.1002/ccd.27196. Epub 2017 Jul 14. PMID 28707316